CLINICAL TRIAL: NCT04393506
Title: Inductive Camrelizumab and Apatinib for Patients With Locally Advanced and Resectable Oral Squamous Cell Carcinoma: A Single-arm Phase I Trial
Brief Title: Inductive Camrelizumab and Apatinib for Patients With Locally Advanced and Resectable Oral Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Icemelting trial
Record Dates: First submitted 2020-05-03; First posted 2020-05-19 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Oral Cancer; VEGFR2 Inhibitor; Programmed Cell Death 1 Inhibitor; Inductive Therapy
MeSH Terms: conditions — Mouth Neoplasms | interventions — camrelizumab; apatinib; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inductive therapy (Other): Inductive therapy with Camrelizumab and Apatinib, followed by radical surgery and post-operative radiotherapy/chemoradiotherapy.
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Procedure: Radical surgery; Radiation: Post-operative radiotherapy/chemoradiotherapy

INTERVENTIONS:
Drug: Camrelizumab — Inductive therapy with Camrelizumab of 200mg, iv, qd, on day 1, 15, 29.
  Other Names: Humanized anti-PD-1 inhibitor
Drug: Apatinib — Inductive therapy with Apatinib of 250mg, po, qd, initiating on day 1, ending on the fifth day before surgery.
  Other Names: VEGFR2 inhibitor
Procedure: Radical surgery — Radical surgery will be performed on the 42th-45th after initiation of inductive therapy
Radiation: Post-operative radiotherapy/chemoradiotherapy — Post-operative radiotherapy/chemoradiotherapy will be performed within 1.5 months after radical surgery, depending on the post-operative pathologic diagnosis.

SUMMARY:
In patients with locally advanced oral squamous cell carcinoma (OSCC), due to the large tumor burden and neck lymph node metastasis, comprehensive treatment is recommended, including surgery, radiotherapy, chemotherapy and others. Pre-operative inductive therapy can reduce tumor volume, increase organ retention rate, and reduce distant metastasis rate. Vascular endothelial growth factor (VEGF) receptor in head and neck squamous cell carcinoma is over-expressed and associated with disease invasion and poor prognosis. The use of targeted therapy against VEGF can not only inhibit tumor neovascularization, but also make the effectiveness of chemotherapeutic agents. VEGF and VEGFR are closely related to immune escape. Tumor growth requires new blood vessels to supply nutrients and oxygen, and VEGF can stimulate neovascularization. However, tumor neovascularization is often abnormal and distorted, which prevents immune active substances from reaching the tumor site. After tumor hypoxia, high expression of VEGF will induce tumor cells to express programmed cell death protein-1 (PD-1), which further leads to immune escape. Targeted drugs against angiogenesis can relieve immunosuppression to a certain extent, and theoretically have a synergistic effect with anti-PD-1 immunotherapy. The innovation of this study is the combination of immune checkpoint inhibitor, Camrelizumab, and targeted drug against VEGFR, Apatinib, as an inductive therapy to treat the patients with locally advanced OSCC, followed with radical surgery and post-operative radiotherapy/chemoradiotherapy, the major pathologic response and safety will be evaluated as the primary surrogate endpoints, the 2-year survival rate and local recurrence rate will be the second endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Eastern cooperative oncology group performance status (ECOG PS) score: 0-2 points
* Pathological diagnosis of oral squamous cell carcinoma (including tongue, gums, cheeks, mouth floor, hard palate, posterior molar region)
* Clinical stage of III/IVA (AJCC 2018)
* Blood routine: white blood cells> 3,000/mm3, hemoglobin> 8g/L, platelets> 80,000/mm3
* Liver function: Alanine Transaminase/Aspartate Transaminase <2.5 times the upper limit of normal, bilirubin <1.5 times the upper limit of normal
* Renal function: serum creatinine <1.5 times the upper limit of normal
* Sign the informed consent

Exclusion Criteria:

* There are still unresolved toxic reactions above CTCAE level 2 caused by previous anti-cancer treatment
* Obvious cardiovascular abnormalities [such as myocardial infarction, superior vena cava syndrome, heart disease of grade 2 or higher diagnosed according to the classification criteria of the New York Heart Association (NYHA) 3 months before enrollment]
* Active severe clinical infection (> CTCAE 5.0 version 2 infection)
* Difficult to control hypertension (systolic blood pressure> 150 mmHg and / or diastolic blood pressure> 90 mmHg) or cardiovascular disease with clinical significance (such as activity)-such as cerebrovascular accident (≤ 6 months before randomization), myocardial infarction (≤6 months before randomization), unstable angina, New York Cardiology Society (NYHA Appendix 5) congestive heart failure grade II or above, or severe arrhythmia that cannot be controlled with drugs or has potential impact on experimental treatment
* Women during pregnancy or lactation
* Participated in other clinical studies within 30 days before enrollment
* Other circumstances that the investigator thinks are not suitable for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Major pathologic response | One year
  Major pathologic response is based on the pathological examination on the post-operative specimens after inductive therapy.

SECONDARY OUTCOMES:
2-year overall survival | Two years
  The overall survival time refers to the time from initiating inductive therapy to death due to any cause.
2-year tumor recurrence rate | Two years
  The tumor recurrence rate is calculated using the number of patients with tumor recurrence divided by the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, PHD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ju WT, Xia RH, Zhu DW, Dou SJ, Zhu GP, Dong MJ, Wang LZ, Sun Q, Zhao TC, Zhou ZH, Liang SY, Huang YY, Tang Y, Wu SC, Xia J, Chen SQ, Bai YZ, Li J, Zhu Q, Zhong LP. A pilot study of neoadjuvant combination of anti-PD-1 camrelizumab and VEGFR2 inhibitor apatinib for locally advanced resectable oral squamous cell carcinoma. Nat Commun. 2022 Sep 14;13(1):5378. doi: 10.1038/s41467-022-33080-8. PMID 36104359

DOCUMENTS (1):
  • Informed Consent Form (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04393506/ICF_000.pdf